CLINICAL TRIAL: NCT05672251
Title: A Phase 2 Study of Loncastuximab Tesirine Plus Mosunetuzumab in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Loncastuximab Tesirine and Mosunetuzumab for the Treatment of Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22414; NCI-2022-10312 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22414 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 3b Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Recurrent Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Biopsy; Specimen Handling; loncastuximab tesirine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (oncastuximab tesirine, mosunetuzumab) (Experimental): Patients receive loncastuximab tesirine IV and mosunetuzumab IV on study. Patients also undergo PET/CT scan, biopsy, and collection of blood samples on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Loncastuximab Tesirine; Biological: Mosunetuzumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Biological: Loncastuximab Tesirine — Given IV
  Other Names: ADC ADCT-402; ADCT-402; Anti-CD19 PBD-conjugate ADCT-402; Loncastuximab Tesirine-lpyl; Zynlonta
Biological: Mosunetuzumab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; Mosunetuzumab-axgb; RG 7828; RG-7828; RG7828; RO7030816
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial studies the safety and how well of loncastuximab tesirine when given together with mosunetuzumab works in treating patients with diffuse large B-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Loncastuximab tesirine is a monoclonal antibody, loncastuximab, linked to a toxic agent called tesirine. Loncastuximab attaches to anti-CD19 cancer cells in a targeted way and delivers tesirine to kill them. Mosunetuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving loncastuximab tesirine with mosunetuzumab may help treat patients with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of loncastuximab tesirine plus mosunetuzumab in patients with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL). (Safety Lead-In) II. Estimate the overall response rate (ORR) in R/R DLBCL patients treated with loncastuximab tesirine plus mosunetuzumab. (Phase 2)

SECONDARY OBJECTIVES:

I. Estimate the complete response (CR) rate, duration of response (DOR), progression-free survival (PFS), and overall survival (OS) in R/R DLBCL patients treated with loncastuximab tesirine plus mosunetuzumab.

II. Evaluate the toxicity of loncastuximab tesirine plus mosunetuzumab for R/R DLBCL.

EXPLORATROY OBJECTIVE:

I. Evaluate genomic and immune biomarkers of response and resistance to loncastuximab tesirine combined with mosunetuzumab

OUTLINE:

Patients receive loncastuximab tesirine intravenously (IV) and mosunetuzumab IV on study. Patients also undergo positron emission tomography (PET)/computed tomography (CT) scan, biopsy, and collection of blood samples on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines.
* Be willing to provide tissue from a fresh core or excisional biopsy (performed as standard of care) of a tumor lesion prior to starting study therapy or from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* Age: >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) =< 2.
* Histologically confirmed diagnosis of diffuse large B-cell lymphoma or Follicular Lymphoma Grade 3B according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution. Subtypes of DLBCL including transformed indolent lymphomas (TIL) including Richter's Transformation, primary mediastinal large B-cell lymphoma (PMBCL), and high-grade B-cell lymphoma not otherwise specified (HGBCL-NOS) are eligible.
* Life expectancy > 12 months.
* Histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma Grade 3B according to the WHO classification, with hematopathology review at the participating institution. Subtypes of DLBCL including transformed indolent lymphomas (TIL) including Richter's Transformation, primary mediastinal large B-cell lymphoma (PMBCL), and high-grade B-cell lymphoma not otherwise specified (HGBCL-NOS) are eligible.
* Relapsed or refractory disease after >= 1 prior line of therapy (prior CD19-directed therapy and prior autologous stem cell transplant are allowed).

  * Relapse at the time of study enrollment must have been confirmed histologically (with hematopathology review at the participating institution). Exceptions may be granted with study PI approval.
* Measurable disease by computerized tomography (CT) or positron emission tomography (PET)/CT scan with one or more sites of disease >= 1.5 cm in longest dimension.
* Tumor must be positive for both CD19 and CD20 by immunohistochemistry after the most recent therapy.
* Fully recovered from the acute toxic effects (except alopecia) to =< Grade 1 to prior anti-cancer therapy
* Without bone marrow involvement: Absolute neutrophil count (ANC) >= 1,000/mm^3.

  * (G-CSF is allowed to reach ANC requirement).
* With bone marrow involvement: no minimum ANC requirement.

  * (G-CSF is allowed to reach ANC requirement).
* Platelets >= 75,000/mm^3.
* Total bilirubin =< 1.5 X upper limit of normal (ULN).

  * If hepatic involvement by lymphoma, or Gilbert's disease: =< 3X ULN.
* Aspartate aminotransferase (AST) =< 2.5 x ULN.

  * If hepatic involvement by lymphoma: AST =< 5 x ULN.
* Alanine aminotransferase (ALT) =< 2.5 x ULN.

  * If hepatic involvement by lymphoma: ALT =< 5 x ULN .
* Creatinine clearance of >= 40 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International Normalized Ratio (INR) OR Prothrombin (PT) =< 1.5 x ULN.
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants.
* If not receiving anticoagulants: Activated Partial Thromboplastin Time (aPTT) =< 1.5 x ULN
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females of childbearing potential to abstain from heterosexual intercourse or use two adequate method of birth control, including at least 1 method with a failure rate of < 1% per year, for at least 28 days prior to Day 1 of Cycle 1, during the treatment period (including periods of treatment interruption), until 3 months after the final dose mosunetuzumab and 9 months after the last dose of loncastuximab tesirine. Women must refrain from donating eggs during this same period. Agreement by males to abstain from heterosexual intercourse or use a condom with female partners of childbearing potential or pregnant female partners during the treatment period and for 3 months after the final dose of mosunetuzumab and 6 months after the last dose of loncastuximab tesirine. Men must refrain from donating sperm during this same period.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only) with no identified cause other than menopause.
  * Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established and proper use of progestogen only hormonal contraceptives that inhibit ovulation, hormone releasing intrauterine devices, and copper intrauterine devices. Barrier methods must always be supplemented with the use of a spermicide. Note: Combined oral contraceptives are not recommended.

Exclusion Criteria:

* Prior treatment with loncastuximab tesirine.
* Prior treatment with mosunetuzumab or other CD20-directed bispecific antibodies.
* Prior allogeneic stem cell transplantation.
* Prior use of any monoclonal antibody, radioimmunoconjugate or ADC within 2 weeks prior to Day 1 of protocol therapy.
* Treatment with any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 2 weeks or 5 half-lives of the drug, whichever is shorter, prior to Day 1 of protocol therapy.
* Treatment with radiotherapy within 2 weeks prior to Day 1 of protocol therapy.

  * If patients have received radiotherapy within 4 weeks prior to prior to Day 1 of protocol therapy, patients must have at least one measurable lesion outside of the radiation field. Patients who have only one measurable lesion that was previously irradiated but subsequently progressed are eligible.
* Autologous stem cell transplantation (SCT) within 30 days prior to prior to Day 1 of protocol therapy.
* Prior treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 30 days prior to Day 1 of protocol therapy.
* Live vaccine within 30 days prior to Day 1 of protocol therapy.
* Concomitant investigational therapy.
* Treatment-emergent immune-related adverse events associated with prior immunotherapeutic agents(e.g., immune checkpoint inhibitor therapies). Note: For certain prior treatments, such as CAR-T cell therapies, patients with prior immune-related Grade >= 3 adverse events (e.g., CRS) may be allowed after discussion with and approval by the Study PI.
* Systemic steroid therapy or any other form of immunosuppressive therapy for lymphoma symptom control must be tapered down to =< 20 mg/day prednisone or equivalent. Exceptions are:

  * Inhaled or topical steroids
  * Use of mineralocorticoids for management of orthostatic hypotension
  * Use of physiologic doses of corticosteroids for management of adrenal insufficiency
* Known hypersensitivity to biopharmaceutical produced in chinese hamster ovary (CHO) cells or history of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents.
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
* History of solid organ transplantation.
* History of progressive multifocal leukoencephalopathy (PML).
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
* Clinically significant uncontrolled illness.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with past HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV deoxyribonucleic acid (DNA) is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). Testing to be done only in patients suspected of having infections or exposures.
* Known active human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable HIV viral load with CD4 > 200 and are on HAART medication are allowed. Testing to be done only in patients suspected of having infections or exposures.
* Known or suspected chronic active Epstein-Barr virus (EBV) infection.
* Known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement.
* History of erythrema multiforme, Grade >= 3 rash, or blistering following prior treatment with immunomodulatory derivatives.
* Symptomatic cardiac disease (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias), cerebrovascular event/stroke or myocardial infarction within the past 6 months.
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis.
* Active autoimmune disease requiring treatment.
* History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with a history of disease-related immune thrombocytopenic purpura, autoimmune hemolytic anemia, or other stable autoimmune diseases may be eligible.
* Recent major surgery (within 4 weeks) prior to start of protocol therapy, other than for diagnosis.
* History of another primary malignancy that has not been in remission for at least 2 years, with the following exceptions:

  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g. cervical, esophageal) without evidence of disease
  * Asymptomatic prostate cancer managed with a watch-and-wait strategy
  * If the malignancy is expected to not require any treatment for at least 2 years (this exception should be discussed with the study PI).
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Unacceptable toxicity (Safety Lead-in) | Up to 30 days post-last dose of protocol therapy
  Defined as any toxicity occurring during the first cycle of treatment for patients enrolled on DL 1, or during the first two cycles of treatment for patients enrolled on DL -1, within at most one out of six patients treated. Will be conducted per the rolling six design.
Overall response rate (ORR) (Phase 2) | Up to 2 years post-last dose
  Defined as the proportion of response-evaluable participants that achieve a best response of either CR or PR. Will use a Simon's 2-stage Minimax design, occur within at most 26 responders. Will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post-last dose of protocol therapy
  Will be graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and cytokine-release syndrome (CRS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading Criteria.
Complete response rate (CR) rate | Up to 2 years post-last dose
  Defined as the proportion of response-evaluable participants that achieve a best response of CR. Will be estimated along with the 95% exact binomial confidence interval.
Duration of response (DOR) | Up to 2 years post-last dose
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Progression-free survival (PFS) | From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier, assessed up to 2 years post-last dose
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Overall Survival (OS) | From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier, assessed up to 2 years post-last dose
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Swetha Kambhampati, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States